CLINICAL TRIAL: NCT03074409
Title: The Modulatory Effect of Oxytocin on Interoception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-34
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Interoception
Keywords: Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): intranasal administration of oxytocin
  Interventions: Drug: oxytocin
- placebo (Placebo Comparator): intranasal administration of the same ingredient except oxytocin
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oxytocin — self-administration of oxytocin (nasal spray)
  Arms: oxytocin
Drug: placebo — self-administration of placebo (nasal spray)
  Arms: placebo

SUMMARY:
This study is designed to investigate oxytocin's effects on interoception and whether these effects vary as a function of different emotional valence.

DETAILED DESCRIPTION:
The present study will use a double-blind, between-subject, placebo-controlled design to investigate the modulatory effect of oxytocin on interoception and whether this effect will vary as a function of emotional valence. In Experiment 1, subjects will perform a heartbeat detection task and the group differences between oxytocin and placebo groups of the interoceptive accuracy and neural activity in the core interoceptive network will be investigated. In Experiment 2, subjects will be asked to watch emotional faces while perform the heartbeat detection task. Investigators will examine whether oxytocin's effects on interoception will be varied as a function of different emotional valence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Subjects reported having any neurological problems, psychiatric illness or drug or alcohol abuse and none were currently taking any form of medication and had not drunk any caffeine-containing beverages on the day of the experiment.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 41 | 42
Completed | 37 | 38
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: 83 subjects were recruited and 8 subjects were excluded due to low quality of electrocardiogram data (6 subjects) or failure of behavioral data acquisition (2 subjects).
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (2.5) | 21.5 (2.4) | 21.35 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 42 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 41 | 42 | 83

OUTCOME MEASURES:

1. Primary Outcome: Heartbeat Detection (Interoception) Accuracy
Description: heartbeat detection (interoception) accuracy is calculated by the following equation: 1/N ∑ (1 - (|recorded heartbeats - counted heartbeats|)/recorded heartbeats). N was the number of blocks for the heartbeat detection task.
Time Frame: 45 minutes after oxytocin/placebo treatment
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: ratio of correct heartbeat counting
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 37 | 38
ratio of correct heartbeat counting | 0.637 (0.035) | 0.735 (0.034)

2. Primary Outcome: Interoceptive Network Activity
Description: interoceptive network (including anterior insula and dorsal cingulate cortex) activity as measured by the functional MRI technique in the heartbeat detection task. In the heartbeat detection task participants were instructed to make a keypress each time they felt their heartbeat. The interoceptive network activity was indicated by the percentage of BOLD signal change. The value of the percentage of BOLD signal change indicates the level of a certain brain region activated (the involvement of a brain region in a specific cognitive process).
Time Frame: 45 minutes after oxytocin/placebo treatment
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: percentage of BOLD signal change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 37 | 38
percentage of BOLD signal change | 0.548 (0.095) | 0.091 (0.092)

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored for 2 weeks after subjects finished the study.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT03074409/Prot_SAP_000.pdf